CLINICAL TRIAL: NCT00064818
Title: Acupuncture Needling on Connective Tissue by Ultrasound
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Other Study IDs: R21AT000300-01 (NIH)
Record Dates: First submitted 2003-07-14; First posted 2003-07-15 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Healthy
Keywords: connective tissue; ultrasound; acupuncture

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to investigate the effect of acupuncture needling on connective tissue using ultrasound techniques both in animals and in humans.

ELIGIBILITY:
* Healthy Humans
* No bleeding disorders
* No anticoagulant therapy
* Cannot be pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46
Dates: Start 2000-09; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Helen M. Langevin, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States